CLINICAL TRIAL: NCT06972290
Title: The Relationship Between Temperament and Menopause Symptoms: A Cross-Sectional Study Using TEMPS-A and MRS Scales
Brief Title: TEMPS-A and Menopause Symptoms
Acronym: TEMPS-MRS
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Cemile ilhan, Principal Investigator, Obstetrics and Gynecology Specialist, Bagcilar Training and Research Hospital
Other Study IDs: 777/28.09.23
Record Dates: First submitted 2025-04-27; First posted 2025-05-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Menopause; Personality; Temperament
Keywords: Menopausal Transition; Personality Traits; Personality Characteristics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates the relationship between temperament traits and menopausal symptoms using the TEMPS-A and MRS scales in women at menopausal transition stages. It is a cross-sectional observational study.

DETAILED DESCRIPTION:
This observational, cross-sectional study aims to investigate the relationship between temperament traits and menopausal symptoms in women in the menopausal transition stage, specifically classified as STRAW stages -1, +1a, and +1b. Participants are recruited from menopause outpatient clinics.

Data are collected through the administration of the validated Temperament Evaluation of Memphis, Pisa, Paris and San Diego Autoquestionnaire (TEMPS-A) and the Menopause Rating Scale (MRS).

Participants voluntarily complete the questionnaires after providing informed consent. All responses are anonymized and securely stored.

Quality assurance measures include verification of data entry, use of validated scales, and compliance with ethical standards approved by the Istanbul Medipol University Non-Interventional Clinical Research Ethics Committee.

No interventions are applied; the study strictly follows observational registry procedures.

ELIGIBILITY:
Inclusion Criteria:

* Women classified as STRAW stages -1, +1a, and +1b (menopausal transition stages)
* Ability to complete questionnaires and provide informed consent

Exclusion Criteria:

* History of hormone therapy during the past 6 months
* History of surgical menopause (bilateral oophorectomy)
* Presence of severe physical disorders (e.g., malignancy, severe cardiovascular diseases)
* Presence of severe psychological disorders (e.g., major depressive disorder, psychosis)

Max Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women in the menopausal transition stage, classified as STRAW stages -1, +1a, and +1b, attending menopause outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
TEMPS-A Depressive Subscale Score at Baseline | Baseline (single time point at enrollment)
  Score from the depressive subscale of the TEMPS-A questionnaire, assessing baseline depressive temperament
TEMPS-A Cyclothymic Subscale Score at Baseline | Baseline (single time point at enrollment)
  Score from the cyclothymic subscale of the TEMPS-A questionnaire, assessing mood instability.
TEMPS-A Hyperthymic Subscale Score at Baseline | Baseline (single time point at enrollment)
  Score from the hyperthymic subscale of the TEMPS-A questionnaire, assessing elevated or overly positive mood tendencies.
TEMPS-A Irritable Subscale Score at Baseline | Baseline (single time point at enrollment)
  Score from the irritable subscale of the TEMPS-A questionnaire, assessing baseline tendency toward irritability.
TEMPS-A Anxious Subscale Score at Baseline | Baseline (single time point at enrollment)
  Score from the anxious subscale of the TEMPS-A questionnaire, assessing trait anxiety.
MRS Somatic Subscale Score at Baseline | Baseline (single time point at enrollment)
  Somatic subscore of the MRS, measuring physical symptoms such as hot flashes and sleep problems.
MRS Psychological Subscale Score at Baseline | Baseline (single time point at enrollment)
  Psychological subscore of the MRS, reflecting symptoms such as depressive mood, irritability, and anxiety.
MRS Urogenital Subscale Score at Baseline | Baseline (single time point at enrollment)
  Urogenital subscore of the MRS, assessing symptoms such as vaginal dryness or urinary complaints.
MRS Total Score at Baseline | Baseline (single time point at enrollment)
  Total score from the Menopause Rating Scale (MRS), reflecting overall menopausal symptom severity.

SECONDARY OUTCOMES:
Correlation Between TEMPS-A Subscale Scores and MRS Total/Subscale Scores | Baseline (single time point at enrollment)
  The relationship between affective temperament traits (TEMPS-A: depressive, cyclothymic, hyperthymic, irritable, and anxious) and menopausal symptom severity (MRS total and subscale scores) will be assessed using Pearson or Spearman correlation coefficients. The analysis aims to determine whether specific temperament profiles are associated with increased symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Cemile Ilhan, MD, Principal Investigator — Bagcilar Training and Research Hospital
Locations (1):
- Bağcılar Training and Reserach Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No